CLINICAL TRIAL: NCT04993911
Title: Effects of Strength and Balance Training to Reduce the Fall Risk in Knee Osteoarthritis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: REC/00849 Mahrukh Hanif
Record Dates: First submitted 2021-08-05; First posted 2021-08-06 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Sports Physical Therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balance training + conventional exercises (Experimental): Assessment will be performed pre and post of intervention. Intervention will be given 3 days a week for 8 weeks. Each session will include a 5-min warm-up on a fitness bike or treadmill before commencement of the program and a 5-min cool period. Participants of this group will receive balance training with conventional treatment. Participants will perform between 2 sets of 5 and 7 repetitions of each exercise.
  Single leg balance
  Walking forward Walking backward Side stepping Walk heel to toe Static exercises with eyes close or open
  CONVENTIONAL EXERCISE PROGRAM :
  TENS for 15 minutes Hot pack for 15 minutes
  Participants will perform between 2 sets of 7 and 10 repetitions of each exercise:
  Quadriceps/hamstring isometric exercises. ROM and active stretching of the hamstring and quadriceps muscle. Active ankle pump. Squats,step-up, sit to stand, calf raises Straigh leg raising exercise in crook lying position
  Interventions: Other: Experimental Group
- Only conventional (Active Comparator): CONVENTIONAL EXERCISE PROGRAM :
  TENS for 15 minutes Hot pack for 15 minutes
  Participants will perform between 2 sets of 7 and 10 repetitions of each exercise:
  Quadriceps/hamstring isometric exercises. ROM and active stretching of the hamstring and quadriceps muscle. Active ankle pump. Squats,step-up, sit to stand, calf raises Straigh leg raising exercise in crook lying position
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Experimental Group — Assessment will be performed pre and post of intervention. Intervention will be given 3 days a week for 8 weeks. Each session will include a 5-min warm-up on a fitness bike or treadmill before commencement of the program and a 5-min cool period. Participants of this group will receive balance training with conventional treatment. Participants will perform between 2 sets of 5 and 7 repetitions of each exercise.
  Single leg balance
  * Walking forward
  * Walking backward
  * Side stepping
  * Walk heel to toe
  * Static exercises with eyes close or open
  CONVENTIONAL EXERCISE PROGRAM :
  * TENS for 15 minutes
  * Hot pack for 15 minutes
  * Participants will perform between 2 sets of 7 and 10 repetitions of each exercise:
  * Quadriceps/hamstring isometric exercises.
  * ROM and active stretching of the hamstring and quadriceps muscle.
  * Active ankle pump.
  * Squats,step-up, sit to stand, calf raises
  * Straigh leg raising exercise in crook lying position
  Arms: Balance training + conventional exercises
Other: Control Group — Participants of this group will receive only conventional therapy which will include; before beginning the program, each session will feature a 5-minute warm-up on a fitness bike or treadmill, followed by a 5-minute cool-down. Participants of this group will receive only conventional therapy which will include.
  * CONVENTIONAL EXERCISE PROGRAM :
  * TENS for 15 minutes
  * Hot pack for 15 minutes
  * Participants will perform between 2 sets of 7 and 10 repetitions of each exercise:
  * Quadriceps/hamstring isometric exercises.
  * ROM and active stretching of the hamstring and quadriceps muscle.
  * Active ankle pump.
  * Squats,step-up, sit to stand, calf raises
  * Straigh leg raising exercise in crook lying position
  Arms: Only conventional

SUMMARY:
This study will address the scarcity of research and the variations in recommendations regarding the effects of strength and balance training to reduce the fall risk in knee osteoarthritis patients.

DETAILED DESCRIPTION:
This Study will be conducted in Alkhidmat Raazi Hospital. Written informed consent for inclusion in the study was taken. Patients of experimental group will receive balance training with conventional along with TENS, heating pad for one hour 3 times weekly. Assessment will be performed pre and post of intervention. Intervention will be given 3 days a week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age from 55 and 80 year
* Both male and female patients.
* Participants will need to have had knee pain for at least 6 months and experience current average pain of at least 3 (on an 11-point Numerical Pain Rating Scale (NRS)
* Patients having no other physical and mental illness.
* Osteoarthritis of knee (Stage-II) by kallgren and lawrence scale

Exclusion Criteria:

* Patients with lab results abnormal (malignancy)
* Nonmusculoskeletal conditions
* Patient's undergone surgery of knee.
* Other than osteoarthritis

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Arthritis Index (WOMAC) | 6-8 Weeks
  It is widely used in the evaluation of Knee Osteoarthritis. It is a questionnaire consisting of 24 items divided into 3 subscales. Pain (5 items), Stiffness (2 items) and Physical Function (17 items). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Numeric rate pain scale | 6-8 Weeks
  This is the scale to measure pain level of participants. is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Berg balance scale (BBS) | 6-8 Weeks
  To measure the functional performance of muscle, balance system. It grade the individual as having high, low and moderate risk of fall. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

CONTACTS AND LOCATIONS:
Overall Officials: Suhail Karim, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Gymnastic physiotherapy and nutrition in bahria town Rawalpindi, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JK, Kim TH, Park SW, Kim HY, Kim Sh, Lee Sy, Lee SM. Protective effects of human placenta extract on cartilage degradation in experimental osteoarthritis. Biol Pharm Bull. 2010;33(6):1004-10. doi: 10.1248/bpb.33.1004. PMID 20522967
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Srikanth VK, Fryer JL, Zhai G, Winzenberg TM, Hosmer D, Jones G. A meta-analysis of sex differences prevalence, incidence and severity of osteoarthritis. Osteoarthritis Cartilage. 2005 Sep;13(9):769-81. doi: 10.1016/j.joca.2005.04.014. PMID 15978850
- [Background] Maly MR. Abnormal and cumulative loading in knee osteoarthritis. Curr Opin Rheumatol. 2008 Sep;20(5):547-52. doi: 10.1097/BOR.0b013e328307f58c. PMID 18698176
- [Background] Kaufman KR, Hughes C, Morrey BF, Morrey M, An KN. Gait characteristics of patients with knee osteoarthritis. J Biomech. 2001 Jul;34(7):907-15. doi: 10.1016/s0021-9290(01)00036-7. PMID 11410174
- [Background] Bennell KL, Hunt MA, Wrigley TV, Hunter DJ, Hinman RS. The effects of hip muscle strengthening on knee load, pain, and function in people with knee osteoarthritis: a protocol for a randomised, single-blind controlled trial. BMC Musculoskelet Disord. 2007 Dec 7;8:121. doi: 10.1186/1471-2474-8-121. PMID 18067658
- [Background] Levinger P, Nagano H, Downie C, Hayes A, Sanders KM, Cicuttini F, Begg R. Biomechanical balance response during induced falls under dual task conditions in people with knee osteoarthritis. Gait Posture. 2016 Jul;48:106-112. doi: 10.1016/j.gaitpost.2016.04.031. Epub 2016 May 6. PMID 27239773
- [Background] Knoop J, Steultjens MP, van der Leeden M, van der Esch M, Thorstensson CA, Roorda LD, Lems WF, Dekker J. Proprioception in knee osteoarthritis: a narrative review. Osteoarthritis Cartilage. 2011 Apr;19(4):381-8. doi: 10.1016/j.joca.2011.01.003. Epub 2011 Jan 18. PMID 21251988
- [Background] Alnahdi AH, Zeni JA, Snyder-Mackler L. Muscle impairments in patients with knee osteoarthritis. Sports Health. 2012 Jul;4(4):284-92. doi: 10.1177/1941738112445726. PMID 23016099
- [Background] Smidt N, de Vet HC, Bouter LM, Dekker J, Arendzen JH, de Bie RA, Bierma-Zeinstra SM, Helders PJ, Keus SH, Kwakkel G, Lenssen T, Oostendorp RA, Ostelo RW, Reijman M, Terwee CB, Theunissen C, Thomas S, van Baar ME, van 't Hul A, van Peppen RP, Verhagen A, van der Windt DA; Exercise Therapy Group. Effectiveness of exercise therapy: a best-evidence summary of systematic reviews. Aust J Physiother. 2005;51(2):71-85. doi: 10.1016/s0004-9514(05)70036-2. PMID 15924510
- [Background] Sherrington C, Tiedemann A, Fairhall N, Close JC, Lord SR. Exercise to prevent falls in older adults: an updated meta-analysis and best practice recommendations. N S W Public Health Bull. 2011 Jun;22(3-4):78-83. doi: 10.1071/NB10056. PMID 21632004
- [Background] Diracoglu D, Aydin R, Baskent A, Celik A. Effects of kinesthesia and balance exercises in knee osteoarthritis. J Clin Rheumatol. 2005 Dec;11(6):303-10. doi: 10.1097/01.rhu.0000191213.37853.3d. PMID 16371799
- [Background] Sharma L, Cahue S, Song J, Hayes K, Pai YC, Dunlop D. Physical functioning over three years in knee osteoarthritis: role of psychosocial, local mechanical, and neuromuscular factors. Arthritis Rheum. 2003 Dec;48(12):3359-70. doi: 10.1002/art.11420. PMID 14673987
- [Background] 14. Aguiar GC, Rocha SG, Rezende GA, Nascimento MR, Scalzo PL. Effects of resistance training in individuals with knee osteoarthritis. Fisioterapia em Movimento. 2016 Sep;29(3):589-96
- [Background] Silva A, Serrao PR, Driusso P, Mattiello SM. The effects of therapeutic exercise on the balance of women with knee osteoarthritis: a systematic review. Rev Bras Fisioter. 2012 Jan-Feb;16(1):1-9. English, Portuguese. PMID 22441221
- [Background] 16. Chhabr HK, Sathya P. Effect of conventional exercises with balance training &only conventional exercises in patients with osteoarthritis of knee. Int J Innov Res Sci Eng. 2015;4(7):5048-6.
- [Background] 17. Efficacy of Balance Training in Combination With Physical Therapy in Rehabilitation of Knee Osteoarthritis: A Randomized Clinical Trial
- [Background] Levinger P, Dunn J, Bifera N, Butson M, Elias G, Hill KD. High-speed resistance training and balance training for people with knee osteoarthritis to reduce falls risk: study protocol for a pilot randomized controlled trial. Trials. 2017 Aug 18;18(1):384. doi: 10.1186/s13063-017-2129-7. PMID 28821271
- [Background] McConnell S, Kolopack P, Davis AM. The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC): a review of its utility and measurement properties. Arthritis Rheum. 2001 Oct;45(5):453-61. doi: 10.1002/1529-0131(200110)45:53.0.co;2-w. No abstract available. PMID 11642645
- [Background] Svensson M, Lind V, Lofgren Harringe M. Measurement of knee joint range of motion with a digital goniometer: A reliability study. Physiother Res Int. 2019 Apr;24(2):e1765. doi: 10.1002/pri.1765. Epub 2018 Dec 27. PMID 30589162
- [Background] Ferraz MB, Quaresma MR, Aquino LR, Atra E, Tugwell P, Goldsmith CH. Reliability of pain scales in the assessment of literate and illiterate patients with rheumatoid arthritis. J Rheumatol. 1990 Aug;17(8):1022-4. PMID 2213777